CLINICAL TRIAL: NCT05612906
Title: Effect of RDN on Renal Function
Brief Title: Renal Nerve Denervation(RDN) and Renal Function
Status: Recruiting | Type: Observational
Sponsor: Zhengrong Huang (Other)
Responsible Party: Sponsor-Investigator, Zhengrong Huang, Professor, The First Affiliated Hospital of Xiamen University
Organization: The First Affiliated Hospital of Xiamen University (Other)
Other Study IDs: 2022-Renal nerve denervation
Record Dates: First submitted 2022-08-18; First posted 2022-11-10 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-07

CONDITIONS: Effects of RDN on Renal Function

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Current studies have found the efficacy of RDN in the treatment of hypertension, however, the safety of RDN in renal function is still lacking. Therefore, the investigators are aimed to study the effect of RDN on renal function.

ELIGIBILITY:
Inclusion Criteria:

1.18<age≤75 years; 2.clinic blood pressure ≥ 140/90 mmHg or 24-hour ambulatory blood pressure monitoring average blood pressure ≥ 135/85 mmHg after taking 3 or more antihypertensive drugs for more than 4 weeks; 3.essential hypertension, renal parenchymal hypertension, or hypertension patients who are willing to receive RDN ; 4.who signed informed consent and were approved by the Ethics Committee of the First Affiliated Hospital of Xiamen University.

Exclusion Criteria:

* pregnant women or lactating patients;

  * identified secondary hypertension or Pseudo hypertension;

    * whose renal arteries were unsuitable for ablation

      * obvious bleeding tendency and blood system diseases;

        * malignant tumors or end-stage diseases; ⑥Severe peripheral vascular disease, abdominal aortic aneurysm; ⑦A history of the acute coronary syndrome within two weeks; ⑧acute or severe systemic infection; ⑨drug or alcohol dependence or refusal to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory hypertension
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes of serum creatinine and urea nitrogen before and after RDN operation | Baseline,1week/1 month/6months after RDN operation
  Serum creatinine(umol/L, ammonia iminohydrolase assay)and urea nitrogen(umol/L, urease methods) were obtained by blood test.
Changes of glomerular filtration rate before and after RDN operation | Baseline, 6months after RDN operation
  Glomerular filtration rate(ml/min) were obtained by ECT

SECONDARY OUTCOMES:
Effect of RDN operation on renal artery | Baseline, 6months after RDN operation
  Renal arteries were observed by CT angiography.
Urinary protein/serum creatinine ratio change before and after RDN operation | Baseline,1week/1 month/6months after RDN operation
  Urinary protein (mg/L, PRM assay) were tested by urine test.Serum creatinine(umol/L, ammonia iminohydrolase assay) were obtained by blood test.

CONTACTS AND LOCATIONS:
Locations (1):
- zhengrong Huang, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided